CLINICAL TRIAL: NCT03526185
Title: A Pilot Study Using Short-Term Cultured Anti-Tumor Autologous Lymphocytes Following a Lymphocyte Depleting Regimen in Metastatic Melanoma
Brief Title: A Pilot Study Using Short-Term Cultured Anti-Tumor Autologous Lymphocytes
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: lack of funds
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Michael Hurwitz, Assistant Professor of Medicine (Medical Oncology), Yale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2000020477
Record Dates: First submitted 2018-01-22; First posted 2018-05-16 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: 2 separate cohorts are included in the study design. These groups will not be directly compared.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): * Subjects will receive a non-myeloablative lymphocyte depleting preparative regimen of cyclophosphamide (60 mg/kg/day IV) on days -7 and -6 and fludarabine (25 mg/m2/day) on days -5 through -1.
  * Prophylactic antibiotics will be administered as medically indicated until recovery of ANC to > 500 and recovery of ALC to > 400
  * On day 0 subjects will receive the infusion of autologous TIL and one hour later (but can be delayed up to 24 hours) will begin low-dose aldesleukin (IL-2) (72,000 IU/kg IV every 12 hours for up to 10 doses).
  Interventions: Drug: Tumor Infiltrating Lymphocytes
- Cohort 2 (Experimental): * Subjects will receive a non-myeloablative lymphocyte depleting preparative regimen of cyclophosphamide (60 mg/kg/day IV) on days -7 and -6 and fludarabine (25 mg/m2/day) on days -5 through -1.
  * Prophylactic antibiotics will be administered as medically indicated until recovery of ANC to > 500 and recovery of ALC to > 400
  * On day 0 subjects will receive the infusion of autologous TIL and one hour later (but can be delayed up to 24 hours) will begin low-dose aldesleukin (IL-2) (72,000 IU/kg IV every 12 hours for up to 10 doses).
  * Within 1 week post discharge subjects will be treated with Nivolumab 1 mg/kg and Ipilimumab 3 mg/kg every 3 weeks for 4 doses. Following this, patients will receive Nivolumab 480 mg every 4 weeks. Adjuvant Nivolumab will continue until evidence of disease progression or inability to tolerate treatment.
  Interventions: Drug: Tumor Infiltrating Lymphocytes; Drug: Nivolumab and Ipilimumab

INTERVENTIONS:
Drug: Tumor Infiltrating Lymphocytes — The regimen consists of treatment with cyclophosphamide and fludarabine,followed by infusion of up to 3x1011 lymphocytes (minimum of 1x109) expanded in vitro from subjects own resected tumor followed by the administration of aldesleukin (IL-2).
  Other Names: Autologous TIL; Unselected TIL; Young TIL
Drug: Nivolumab and Ipilimumab — • Within 1 week post discharge subjects will be treated with Nivolumab 1 mg/kg and Ipilimumab 3 mg/kg every 3 weeks for 4 doses. Following this, patients will receive Nivolumab 480 mg every 4 weeks. Adjuvant Nivolumab will continue until evidence of disease progression or inability to tolerate treatment.
  Arms: Cohort 2

SUMMARY:
To determine the feasibility and safety of administering a regimen of TIL/IL-2, using a cell product manufactured in the Yale Advanced Cell Therapy Laboratories, in subjects with metastatic melanoma who are not responding or have progressed after receiving prior therapy with a PD-1/PD-L1 antagonist used alone or in combination with anti-CTLA-4. Additionally, a second cohort of patients with metastatic melanoma who are not responding or have progressed after receiving prior therapy with a PD-1/PD-L1 antagonist alone or in combination with anti-CTLA-4 will receive anti-PD-1 and anti-CTLA-4 therapy with Nivolumab and Ipilimumab.

DETAILED DESCRIPTION:
The objectives of this study have been expanded since its original registration to inlcude an additional cohort of patients (now designated Cohort 1 and Cohort 2). Cohort 1 is the original group of patients described in the initial registration of the study.

Cohort 1 Objectives:

* To determine the feasibility and safety of administering a regimen of TIL/IL-2, using a cell product manufactured in the Yale Advanced Cell Therapy Laboratories, in subjects with metastatic melanoma who are not responding or have progressed after receiving prior therapy with a PD-1/PD-L1 antagonist used alone or in combination with anti-CTLA-4.
* To assess for evidence of clinical activity.
* To conduct a preliminary assessment of the TCR clonotypes present in marker positive CD8+ cells (4-1BB, LAG-3, TIM-3, PD-1) versus marker-negative CD8+ T-cells early in the expansion cultures and compare to clonotypes late in the final product and in peripheral blood lymphocytes (PBL) 1 and 2 months post infusion.

Cohort 2 Objectives:

* To determine the feasibility and safety of administering a regimen of TIL/IL-2, using a cell product manufactured in the Yale Advanced Cell Therapy Laboratories, followed by anti-PD-1 and anti-CTLA-4 therapy with Nivolumab and Ipilimumab in subjects with metastatic melanoma who are not responding or have progressed after receiving prior therapy with a PD-1/PD-L1 antagonist alone or in combination with anti-CTLA-4.
* To evaluate the efficacy of TIL/IL-2 therapy in combination with subsequent anti-PD-1 Nivolumab and anti-CTLA-4 Ipilimumab by assessing the objective response rate by immune-related RECIST (irRECIST).
* To conduct a preliminary assessment of the TCR clonotypes present in marker positive CD8+ cells (e.g. 4-1BB, LAG-3, TIM-3, PD-1) versus marker-negative CD8+ T-cells early in the expansion cultures and compare to clonotypes late in the final product and in peripheral blood lymphocytes (PBL) 1 and 2 months post infusion.

ELIGIBILITY:
Inclusion Criteria:

For Cohorts 1 and 2:

* Metastatic melanoma;
* A metastatic lesion at least 1.5 cm in diameter that can be removed surgically
* Measurable or evaluable disease not including the resected lesion
* ECOG PS of 0 or 1 prior to cell harvest
* Assessment by the treating physician that ECOG performance status of no higher than 2 can be maintained at least for the period of cell generation, lymphoablation, cell infusion and IL-2 administration (for at least 6 weeks following cell harvest)
* Tumor refractory to or progressing following prior PD-1/PD-L1 therapy alone or in combination with an anti-CTLA-4 agent
* Ability to understand risks and benefits of the treatment and to give informed consent

Exclusion Criteria:

For Cohorts 1 and 2:

* Received prior cell transfer therapy that included non-myeloablative or ablative chemotherapy
* Any significant major organ dysfunction (see protocol)
* Residual toxicity > gr1 from immune checkpoint inhibitor other than persistent endocrinopathy on hormone replacement; all symptoms of prior colitis and enteritis must have resolved completely as assessed by history
* Any contraindication to neutropenia or thrombocytopenia for up to 2 weeks (no active major infection, no site of active, clinically significant bleeding)
* Concurrent major medical illnesses
* Any form of immunodeficiency
* Requirement for steroids > 10 mg prednisone daily or equivalent
* Severe hypersensitivity to any of the agents used in this study
* Contraindications for IL-2 administration

At the time of lymphoablation subjects must meet baseline eligibility criteria with the following additions and exceptions:

• Confirmation by lab that cell product can be ready for harvest and infusion within 7 days

For Cohort 2 only:

At the time of the start of anti-PD-1/anti-CTLA-4 therapy, subjects must meet baseline eligibility criteria with the following additions and exceptions:

* Patient cannot have a steroid requirement > 10 mg prednisone daily or equivalent
* Patients who have received prior PD-1/PD-L1 antagonist therapy and developed severe autoimmune disease precluding further immune checkpoint therapy
* Any organ dysfunction that makes the subject ineligible for anti-PD1 and anti-CTLA-4 treatment as deemed by the treating investigator
* ECOG PS of 0-2
* Hgb of at least 8.0 gm/dl (may be transfused to this level)
* Creatinine not greater than 2.5 mg/dl
* AST or ALT not > 5x ULN and total bilirubin not > 2.5 mg/dl
* No clinically significant change in major organ function compared to initial eligibility evaluation
* Prior to initiating the lymphoablation regimen, there can be no untreated brain lesion > 1.0 cm, and/or with significant evidence of hemorrhage. Subjects may begin lymphoablation no less than 1 full day after completing WBRT or stereotactic radiotherapy for brain lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Adverse Events | up to 12 months
  To determine the safety of administering a regimen of TIL/IL-2, incidence of drug-related adverse events (AEs) will be summarized across adverse event type in terms of frequency by event type.
Serious Adverse Events | up to 12 months
  To determine the safety of administering a regimen of TIL/IL-2, serious adverse events (SAEs) will be summarized across event type in terms of frequency by event type. SAE's will include events leading to discontinuation, deaths and clinical laboratory test abnormalities

SECONDARY OUTCOMES:
Objective response rate to TIL | up to 12 months
  Objective response rate (ORR) of the TIL/IL-2 regimen based on investigator review of radiographic images using RECIST 1.1 criteria

OTHER OUTCOMES:
Assessment of Immune features of TIL: 4-1BB | up to 12 months
  to conduct a preliminary assessment of TCR clonotypes using deep sequencing of TCRs from the cell product and of immunologic markers present in marker positive CD8+ cells (specifically 4-1BB, LAG-3, TIM-3, PD-1)
Assessment of Immune features of TIL: LAG-3 | up to 12 months
  to conduct a preliminary assessment of TCR clonotypes using deep sequencing of TCRs from the cell product and of immunologic markers present in marker positive CD8+ cells (specifically 4-1BB, LAG-3, TIM-3, PD-1)
Assessment of Immune features of TIL: TIM-3 | up to 12 months
  to conduct a preliminary assessment of TCR clonotypes using deep sequencing of TCRs from the cell product and of immunologic markers present in marker positive CD8+ cells (specifically 4-1BB, LAG-3, TIM-3, PD-1)
Assessment of Immune features of TIL: PD-1 | up to 12 months
  to conduct a preliminary assessment of TCR clonotypes using deep sequencing of TCRs from the cell product and of immunologic markers present in marker positive CD8+ cells (specifically 4-1BB, LAG-3, TIM-3, PD-1)

CONTACTS AND LOCATIONS:
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States